CLINICAL TRIAL: NCT07119398
Title: Combination Oxytocin/Foley Versus Oxytocin Alone for Induction of Labor in Patients With Preterm Prelabor Rupture of Membranes
Brief Title: Oxytocin/Foley vs. Oxytocin for Induction in Patients With PPROM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Marwan Ma'ayeh, Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-04-FB-0086
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Preterm PROM (Pregnancy)
Keywords: Induction; PPROM; Preterm prelabor rupture of membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: This study is a non-blinded prospective randomized pilot trial of pregnant patients with a singleton pregnancy between 34 weeks 0 days and 36 weeks 6 days gestation with PPROM receiving an induction of labor. Participants will be randomized to either:
  * Induction of labor with intravenous oxytocin
  * Induction of labor with intravenous oxytocin and a transcervical Foley catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin plus Foley (Experimental): • Induction of labor with intravenous oxytocin and a transcervical Foley catheter
  Interventions: Combination Product: Oxytocin plus Foley Catheter
- Oxytocin Only (Active Comparator): • Induction of labor with intravenous oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Combination Product: Oxytocin plus Foley Catheter — Intravenous oxytocin and a transcervical Foley catheter
  Arms: Oxytocin plus Foley
Drug: Oxytocin — Intravenous oxytocin
  Arms: Oxytocin Only

SUMMARY:
Data on the optimal mode of labor induction after preterm prelabor rupture of membranes (PPROM) is lacking. Studies have shown no difference between oxytocin and misoprostol use for labor induction in this cohort (1). The preponderance of evidence from term pregnancies suggests that Foley catheter coupled with oxytocin is better than oxytocin alone, with a higher rate of delivery within 24 hours when a Foley catheter followed by oxytocin is compared to oxytocin alone. However, the use of a Foley catheter has not been evaluated in prospective studies on patients with PPROM.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-50 years of age;
* The patient is fluent in English, physically and mentally able to understand the informed consent, and is willing to participate in this study;
* PPROM;
* Cervical dilation </= 2cm
* Fetal cephalic presentation;
* The patient is between 34 weeks 0 days and 36 weeks 6 days of gestation at the time of enrollment. Gestational age will be determined by last menstrual period, confirmed with a first trimester ultrasound, per the recommended guidelines by the American College of Obstetricians and Gynecologists.

Exclusion Criteria:

* Spontaneous labor
* Known allergy to latex;
* Cervical dilation >2cm;
* Chorioamnionitis;
* Contraindications to induction of labor or use of Foley for cervical ripening
* HIV
* Known or suspected fetal anomaly or aneuploidy;
* Prisoners.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Vaginal Delivery within 12 Hours | 12 hours
  Vaginal Delivery within 12 hours of induction

SECONDARY OUTCOMES:
Vaginal Delivery Rate | From enrollment until delivery
  Overall vaginal delivery rate
Intraamniotic Infection | Enrollment through 6 weeks postpartum
Operative vaginal delivery | From enrollment until delivery
Cesarean delivery | From enrollment until delivery
Estimated and quantitative blood loss | From enrollment until hospital discharge (up to 5 days post-delivery).
Blood transfusion | From enrollment until hospital discharge (up to 5 days post-delivery)
Maternal morbidity and adverse maternal outcomes | From enrollment until 6 weeks postpartum
  Including endometritis / chorioamnionitis, wound infection, venous thromboembolism, massive transfusion and postpartum hemorrhage, ICU admission, and maternal death
Antepartum, intrapartum, or neonatal death | From enrollment until 6 weeks postpartum
Suspected and confirmed neonatal sepsis | From delivery until hospital discharge (up to 5 days post-delivery)
Birth weight | Recorded day of delivery
Hypoglycemia (glucose < 35 mg/dl) requiring IV glucose therapy | From birth until hospital discharge (up to 5 days post-delivery)
Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiopulmonary resuscitation within first 72 hours | From birth until 72 hours after delivery
Neonatal encephalopathy | From birth until hospital discharge (up to 5 days after delivery)
  As defined by the NICHD Neonatal Research Network criteria
Seizures | From birth until hospital discharge (up to 5 days post-delivery)
Shoulder dystocia | Recorded day of delivery
Birth trauma | Recorded day of delivery
  Bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage, or facial nerve palsy
Intracranial hemorrhage | From birth until hospital discharge (up to 5 days post-delivery)
  Intraventricular hemorrhage, subgaleal hematoma, subdural hematoma, or subarachnoid hematoma
Hyperbilirubinemia requiring phototherapy or exchange transfusion | From birth until hospital discharge (up to 5 days post-delivery)
NICU admission | From birth until time of NICU admission or hospital discharge (up to 5 days post-delivery), whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Ma'ayeh, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- [Background] Gomez Slagle HB, Hoffman MK, Sciscione AC, Ma'ayeh M. Combination Foley Catheter-Oxytocin versus Oxytocin Alone following Preterm Premature Rupture of Membranes. Am J Perinatol. 2024 May;41(S 01):e3030-e3034. doi: 10.1055/a-2185-4102. Epub 2023 Oct 4. PMID 37793430
- [Background] Amorosa JMH, Stone J, Factor SH, Booker W, Newland M, Bianco A. A randomized trial of Foley Bulb for Labor Induction in Premature Rupture of Membranes in Nulliparas (FLIP). Am J Obstet Gynecol. 2017 Sep;217(3):360.e1-360.e7. doi: 10.1016/j.ajog.2017.04.038. Epub 2017 May 4. PMID 28479288
- [Background] Mackeen AD, Durie DE, Lin M, Huls CK, Qureshey E, Paglia MJ, Sun H, Sciscione A. Foley Plus Oxytocin Compared With Oxytocin for Induction After Membrane Rupture: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):4-11. doi: 10.1097/AOG.0000000000002374. PMID 29215519
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Schoen CN, Grant G, Berghella V, Hoffman MK, Sciscione A. Intracervical Foley Catheter With and Without Oxytocin for Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jun;129(6):1046-1053. doi: 10.1097/AOG.0000000000002032. PMID 28486381
- [Background] Lin MG, Nuthalapaty FS, Carver AR, Case AS, Ramsey PS. Misoprostol for labor induction in women with term premature rupture of membranes: a meta-analysis. Obstet Gynecol. 2005 Sep;106(3):593-601. doi: 10.1097/01.AOG.0000172425.56840.57. PMID 16135593

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT07119398/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT07119398/ICF_001.pdf